CLINICAL TRIAL: NCT04199143
Title: Cerebrovascular Reactivity to Nitrous Oxyde in Resistant Depression: the PROTOBRAIN Pilote Study
Brief Title: Brain Reactivity to Nitrous Oxyde in Depression : an MRI and Ultrasound Study (PROTOBRAIN Pilote)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DR190058
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression; Nitrous Oxyde
Keywords: Magnetic Resonance Imaging; Ultrasound; Tissue Pulsatility Imaging; Treatment Resistant Depression; Nitrous Oxyde
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — kalinox; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Open-label, Longitudinal, Monocentric, Physiological study comparing depressive patients (responders versus non-respondeurs to Nitrous Oxyde) and healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy voluntary controls (Experimental): A single Non-blinded One-hour administration of 50% Nitrous oxyde (N2O) 50%oxygen (O2) Gas Mixture
  Interventions: Drug: Nitrous Oxide-Oxygen; Device: Tissue Pulsatility Imaging - TPI; Device: Magnetic Resonance Imaging - MRI
- Depressive Patients (Experimental): A single Non-blinded One-hour administration of 50% Nitrous oxyde (N2O) 50%oxygen (O2) Gas Mixture
  Interventions: Drug: Nitrous Oxide-Oxygen; Device: Tissue Pulsatility Imaging - TPI; Device: Magnetic Resonance Imaging - MRI

INTERVENTIONS:
Drug: Nitrous Oxide-Oxygen — The medical product used in this study is a gas for common medical use in various domains including anesthesic, consisting in the equimolar mixture of nitrous oxide and oxygen. Subjects will receive a mixture of 50% N2O / 50% O2 for 1 hour.
  Other Names: KALINOX® 50 %/50 %
Device: Tissue Pulsatility Imaging - TPI — Tissue Pulsatility Imaging (TPI) is a variation of ultrasonic Doppler strain imaging we are developing to measure the local expansion and relaxation of the brain tissue over the cardiac cycle to characterize and image perfusion.
Device: Magnetic Resonance Imaging - MRI — Structural and Functionnal (including BOLD and ASL) MRI will be aquired in this study

SUMMARY:
Recent evidence suggest that Nitrous Oxyde (N2O) could exhibit antidepressant effect in treatment-resistant depression (TRD). However, the pathophysiology of this effect remains unclear and could include glutamatergic activity but also cerebrovascular effects and changes in brain connectivity. The goal of our study is to characterize brain reactivity to N2O in TRD patients, as assessed with Ultrasound Tissue Pulsatility Imaging (TPI) and Magnetic Resonance Imaging (MRI) (including Arterial Spin Labeling - ASL - for brain perfusion and Blood-Oxygen-Level Dependent - BOLD - for brain connectivity and pulsatility).

Ultrasound and MRI Neuroimaging will be measured before, during and after a single one-hour exposure of a 50%N20/50%O2 mixture, in depressed individuals (n=20) and healthy volunteers (n=10). We make the hypothesis that brain reactivity will be lower in depressed individuals nonresponders to N2O compared to responders and healthy controls. This study would provide further characterisation of the pathophysiology of the antidepressant response to N2O, as well as providing potential biomakers (Ultrasound and MRI) for treatment response to N2O in TRD.

DETAILED DESCRIPTION:
Neuroimaging examinations will include:

* Ultrasound Tissue Pulsatility Imaging for assessment of Brain Tissue Pulsatility (BTP) which reflects reactivity in brain movements and mechanical brain properties
* MRI with structural and functional assessments, namely brain volumes, white matter lesions, ASL for brain perfusion and BOLD for resting-state connectivity and brain pulsatility

MRI will be performed before and after a single one-hour exposure of 50%N2O/50%O2 mixture. Ultrasound will be performed before, after and also during gas exposure. Changes in these neuroimaging parameters will constitute the primary assessment of the study. Psychometric and safety assessements will complete the neuroimaging outcomes.

Follow-up will includes 1) a baseline visit for baseline MRI and Psychometric assessements, 2) a second visit for gas exposure and neuroimaging assessements, 3) a third and fourth visits for psychometric and safety assessements, respectively 24 hours and one week after gas exposure.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria common to all participants
* Female between 25 and 50 years of age
* A person who can undergo N2O diffusion via a facial mask.
* A person who has signed an informed consent.
* Person affiliated with a social security scheme.
* Inclusion Criteria for Depressive Patients
* Major Depressive Episode according to DSM-5 criteria, confirmed by the MINI - International Neuropsychiatric Interview.
* Patients with an MADRS score greater than 20 (Montgomery
* Asberg Depression Rating Scale).
* Patients resistant to at least one well-conducted antidepressant treatment, as documented by the MGH-ATRQ scale.
* Absence of: bipolar disorder, schizophrenic disorder, neurodegenerative disease, schizophrenic disorder, neurodegenerative disease, addiction to one or more toxics documented by the MINI.
* Inclusion criteria for healthy voluntary controls
* Absence of: bipolar disorder, schizophrenic disorder, neurodegenerative disease, schizophrenic disorder, neurodegenerative disease, addiction to one or more toxics documented by the MINI, current or past.

Exclusion Criteria:

* Unstable somatic pathology (including unstable neurological or cardiological pathologies at risk of interfering with N2O diffusion)
* Presence of active and significant psychotic symptoms, at investigator's discretion
* Contraindications to mixture 50%N2O/ 50%O2: intracranial hypertension, altered state of consciousness, head trauma, pneumothorax, emphysema bubbles, abdominal gaseous distension, administration of less than 3 months of ophthalmic gas (SF6, C3F8,C2F6) used in eye surgery, known and unsubstituted deficiency in vitamin B12 or folic acid, recent and unexplained neurological abnormalities.
* Contraindications to MRI, including claustrophobia.
* Female who is pregnant or breastfeeding or able to procreate without an effective contraceptive method
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, purpose or consequences of the study (including major under legal protection).
* A person participating in a drug clinical trial or during a period of exclusion from any clinical study due to previous involvement.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Brain Tissue Pulsatility (BTP) as measured with Ultrasound TPI | 3 months after LVLS
  BTP will be measured before, during and after N2O exposure

SECONDARY OUTCOMES:
Brain Volumes (MRI) | 6 months after LVLS
White Matter Lesions (MRI) | 6 months after LVLS
Resting-State Connectivity (BOLD-MRI) | 6 months after LVLS
Brain Pulsatility (BOLD-MRI) | 6 months after LVLS
Brain Perfusion in Arterial Spin Labelling (ASL-MRI) | 6 months after LVLS
Hamilton scale for depression, 17-items | 6 months after LVLS
POMS - Profile of Mood State | 6 months after LVLS
QIDS-SR - Quick Inventory of depressive Symptomatology Self Report | 6 months after LVLS
CGI - Clinical Global Impressions | 6 months after LVLS
STAI-Y-A - State-Trait Anxiety Inventory | 6 months after LVLS
subjective VAE- Visual Analog Evaluation | 6 months after LVLS
SSI - Scale for Suicidal Ideation | 6 months after LVLS
YMRS - Young Mania Rating Scale | 6 months after LVLS
CADSS - Clinician administered dissociative States | 6 months after LVLS
BPRS - Brief Psychiatric Rating Scale | 6 months after LVLS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas DESMIDT, Principal Investigator — CHRU de TOURS
Locations (1):
- University Hospital of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Desmidt T, Dujardin PA, Andersson F, Brizard B, Remenieras JP, Gissot V, Arlicot N, Barantin L, Espitalier F, Belzung C, Tanti A, Robert G, Bulteau S, Gallet Q, Kazour F, Cognet S, Camus V, El-Hage W, Poupin P, Karim HT. Changes in cerebral connectivity and brain tissue pulsations with the antidepressant response to an equimolar mixture of oxygen and nitrous oxide: an MRI and ultrasound study. Mol Psychiatry. 2023 Sep;28(9):3900-3908. doi: 10.1038/s41380-023-02217-6. Epub 2023 Aug 17. PMID 37592013